CLINICAL TRIAL: NCT00068237
Title: A Phase II Study Of Submandibular Salivary Gland Transfer To The Submental Space Prior To Start Of Radiation Treatment For Prevention Of Radiation-Induced Xerostomia In Head And Neck Cancer Patients
Brief Title: Salivary Gland Surgery Before Radiation Therapy in Preventing Radiation-Caused Xerostomia in Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RTOG-0244; CDR0000287213
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2014-01-31 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Head and Neck Cancer; Radiation Toxicity; Xerostomia
Keywords: xerostomia; radiation toxicity; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; untreated metastatic squamous neck cancer with occult primary; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries; Xerostomia; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgery + Transfer + Radiation (Experimental): Submandibular salivary gland transfer at the time of surgery for the primary tumor and neck nodes followed by post-operative radiation therapy.
  Interventions: Procedure: salivary gland transfer; Radiation: Post-operative radiation therapy

INTERVENTIONS:
Procedure: salivary gland transfer — Seikaly and Jha method of submandibular salivary gland transfer at the time of surgery for the primary tumor and neck nodes on Day 1
Radiation: Post-operative radiation therapy — Dose ranging from 54-70 Gy over 5.5-7 weeks, at 2.0 Gy/fraction. Starts within 4-6 weeks of surgery.

SUMMARY:
RATIONALE: Moving a salivary gland out of the area that will undergo radiation therapy may protect the gland from side effects of radiation therapy and may prevent xerostomia (dry mouth).

PURPOSE: Phase II trial to study the effectiveness of salivary gland surgery in preventing xerostomia in patients who are undergoing radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the reproducibility of the surgical technique of submandibular salivary gland transfer in patients with head and neck cancer.
* Determine the rate and severity of radiation-induced xerostomia after this surgery in these patients.
* Determine the pattern of recurrence, disease-free survival, and overall survival of patients treated with this surgery followed by radiotherapy.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients undergo surgical transfer of the submandibular salivary gland to the submental space.

Within 4-6 weeks after surgery, patients undergo radiotherapy once daily, 5 days a week for 5 ½ to 7 weeks in the absence of disease progression or unacceptable toxicity.

Salivary scans are performed before surgery, at 2-3 weeks after surgery, and then at 6 months from the start of radiotherapy.

Quality of life is assessed at baseline and at 3, 6, and 12 months from the start of radiotherapy.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years and then annually.

PROJECTED ACCRUAL: A total of 11-48 patients will be accrued for this study within 1.6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Histologically confirmed, previously untreated squamous cell carcinoma of the oropharynx, hypopharynx, or larynx
  * Head and neck cancer of unknown primary with unilateral metastases to the neck nodes
* No N3 disease
* No carcinoma of the oral cavity or nasopharynx
* No bilateral neck node involvement
* No suspicious neck node on the contralateral neck or the side chosen for salivary gland transfer by CT scan or MRI
* No pre-epiglottic space involvement
* No involvement of level 1 nodes on either side of the neck
* No salivary gland malignancy
* No recurrent disease

PATIENT CHARACTERISTICS:

Age

* At least 18 years old

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin at least 10 g/dL

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No salivary gland disease (e.g., Sjögren's syndrome)
* No other malignancy within the past 3 years except basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 3 years since prior chemotherapy
* No prior or concurrent neoadjuvant chemotherapy
* Concurrent adjuvant chemoradiotherapy (in addition to study radiotherapy) allowed

Endocrine therapy

* Not specified

Radiotherapy

* See Chemotherapy
* No prior radiotherapy to the head and neck
* No concurrent intensity-modulated radiotherapy

Surgery

* Not specified

Other

* No concurrent cholinergic drugs
* No concurrent anti-cholinergic drugs
* No concurrent tricyclic drugs
* No concurrent prophylactic amifostine or pilocarpine during and for at least 3 months after completion of study radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2003-08; Primary Completion 2008-01 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naresh Jha, MBBS, Study Chair — Cross Cancer Institute at University of Alberta
Locations (12):
- United States (9):
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
- Canada (3):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec

REFERENCES:
- [Result] Jha N, Harris J, Seikaly H, Jacobs JR, McEwan AJ, Robbins KT, Grecula J, Sharma AK, Ang KK. A phase II study of submandibular gland transfer prior to radiation for prevention of radiation-induced xerostomia in head-and-neck cancer (RTOG 0244). Int J Radiat Oncol Biol Phys. 2012 Oct 1;84(2):437-42. doi: 10.1016/j.ijrobp.2012.02.034. Epub 2012 Apr 27. PMID 22541957

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgery + Transfer + Radiation
Started | 49
Completed | 44 (Subjects contributing data to the primary analysis are considered to have completed the study.)
Not Completed | 5
Not completed — Ineligible | 3
Not completed — No protocol treatment received | 2

BASELINE CHARACTERISTICS:
Population: All eligible patients who started study treatment.
Arm/Group | Surgery + Transfer + Radiation
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 56.5 [42 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Scored as Having the Surgical Technique of Submandibular Salivary Gland Transfer Performed "Per Protocol"
Description: Surgery will be scored as "per protocol prescription" if scored as such by both central reviewers- the Study Chair and the Radiation Therapy Oncology Group Head and Neck Committee Surgical Chair. If 21 or more of 43 subjects are scored as having surgery "per protocol prescription", then the technique will be considered reproducible with 80% power and 5% type I error using Simon's two stage design with unacceptable/acceptable rates set at 60%/80%.
Time Frame: At the time of the submandibular salivary gland transfer
Population: Eligible patients who started study treatment.
Measure: Number; unit: participants
Arm/Group | Surgery + Transfer + Radiation
Number analyzed (Participants) | 44
participants | 34

2. Secondary Outcome: Percentage of Patients With Acute Xerostomia
Description: The proportion of patients who experience grade 2 or higher xerostomia or start amifostine and/or pilocarpine within 90 days of the start of radiation therapy. A proportion less than or equal to 51% would be considered acceptable based on the results of the U.S. Bioscience phase III amifostine trial (this trial preceded FDAAA requirements).
Time Frame: From start of treatment to 90 days
Population: Eligible patients who started RT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery + Transfer + Radiation
Number analyzed (Participants) | 43
percentage of participants | 25.6 [12.5 to 38.6]

3. Secondary Outcome: Percentage of Patients With Normal Functioning Transferred Submandibular Gland
Description: Salivary gland functioning classified as "Non-functioning", "Minimal function", "Well-functioning but some impairment", "Normal functioning", or "Other" is determined by central review of scintigraphy scans using sodium pertechnetate (Na-99mTcO4-) with a sialagogue (lemon juice) administered halfway through the study to determine if secretory function is maintained.
Time Frame: Pre-surgery, post-surgery (4-6 weeks), post radiation therapy (10-13 weeks)
Population: Eligible patients with salivary scans submitted
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery + Transfer + Radiation
Number analyzed (Participants) | 37
percentage of participants
  Pre-surgery | 70.3 [55.5 to 85.0]
  Post-surgery: number analyzed (Participants) | 36
  Post-surgery | 16.7 [4.5 to 28.8]
  Post-radiotherapy: number analyzed (Participants) | 27
  Post-radiotherapy | 0.0 [0.0 to 0.0]

4. Secondary Outcome: Change From Baseline to One Year in Total Score on the Modified University of Washington Head and Neck Symptom Questionnaire
Description: The University of Washington Head and Neck Symptom Questionnaire, also referred to as the University of Washington Health Related Quality of Life tool (UW-QOL) was modified for use by the Radiation Therapy Oncology Group (RTOG). The resulting UW-QOL-RTOG modification is a valid tool that can be used to assess symptom burden of head and neck cancer patients receiving radiation therapy or those who have recently completed radiation. The UW-QOL-RTOG modification consists of 15 items with response options ranging from 10-50, in multiples of 10. That is, the lowest symptom burden is rated as 10, while the highest symptom burden is rated as 50. The individual item scores are averaged to obtain the final score which also ranges from 10 to 50. This scoring results in a lower score indicating greater HR-QOL; and conversely, higher scores indicating lower health-related quality of life (HR-QOL). Change = baseline score - one year score, such that a positive change score indicates improvement.
Time Frame: Baseline and one year
Population: Eligible patients with both baseline and 1-year questionnaire completed
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Surgery + Transfer + Radiation
Number analyzed (Participants) | 22
score on a scale | 13.6 [7.7 to 16.5]

5. Secondary Outcome: Percentage of Patients Experiencing Facial Edema Following Surgery
Description: Facial edema was noted as present or absent following surgery.
Time Frame: From surgery to 30 days after surgery
Population: Eligible patients who received the procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery + Transfer + Radiation
Number analyzed (Participants) | 44
percentage of participants | 13.6 [3.5 to 23.8]

6. Secondary Outcome: Percentage of Patients Experiencing Acute Grade 3-4 Toxicity Definitely, Probably, or Possibly Related to Radiation Therapy or Chemotherapy
Description: Adverse events are graded using the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) v2.0. Grade refers to the severity of the toxicity by assigning Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to toxicity. "Acute" refers to toxicities occurring less than or equal to 90 days from the start of radiation therapy.
Time Frame: From start of radiation therapy to 90 days
Population: Eligible patients who started RT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery + Transfer + Radiation
Number analyzed (Participants) | 43
percentage of participants | 34.9 [20.6 to 49.1]

7. Secondary Outcome: Percentage of Patients Experiencing Late Grade 3-4 Toxicity Definitely, Probably, or Possibly Related to Radiation Therapy
Description: Adverse events are graded using the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) v2.0. Grade refers to the severity of the toxicity by assigning Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to toxicity. "Late" refers to toxicities occurring at least 91 days from the start of radiation therapy.
Time Frame: From 91 days from start of radiation therapy to last follow-up. Maximum follow-up at time of analysis was 5.6 years.
Population: Eligible patients who started RT and had toxicity data at least 90 days from the end of RT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery + Transfer + Radiation
Number analyzed (Participants) | 38
percentage of participants | 7.9 [0.0 to 16.5]

8. Secondary Outcome: Disease-free Survival Rate at 2 Years
Description: Failure was defined as local, regional, or distant recurrence/progression, second primary tumor, or death due to any cause. Disease-free survival time is defined as time from registration to the the date of failure or last known follow-up (censored). Disease-free survival rate is estimated using the kaplan-meier method.
Time Frame: From registration to two years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery + Transfer + Radiation
Number analyzed (Participants) | 44
percentage of participants | 71.7 [58.2 to 85.3]

9. Secondary Outcome: Overall Survival Rate at 2 Years
Description: Failure was defined as death due to any cause. Survival time is defined as time from registration to the the date of failure or last known follow-up (censored). Survival rate is estimated using the kaplan-meier method.
Time Frame: From registration to two years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgery + Transfer + Radiation
Number analyzed (Participants) | 44
percentage of participants | 76.4 [63.6 to 89.2]

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-SAE adverse events (AE). Please note that different numbers of patients were at risk for different treatment-specific adverse events due to the timing and sequence of treatments.
Arm/Group | Surgery + Transfer + Radiation
Serious Adverse Events (participants affected / at risk) | 2/44
Other Adverse Events (participants affected / at risk) | 38/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Surgery + Transfer + Radiation (N=44)
Anorexia (Metabolism and nutrition disorders) | 1/43
Confusion (Psychiatric disorders) | 1/43
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1/43
Acute Surgical Complication: Bleeding/hematoma (Surgical and medical procedures) | 2
Acute Surgical Complication: Cerebral embolism/CVA (Surgical and medical procedures) | 1
Acute Surgical Complication: Wound infection (Surgical and medical procedures) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Surgery + Transfer + Radiation (N=44)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4/43
Lymphatics-Other (Blood and lymphatic system disorders) | 1/43
Hearing impaired (Ear and labyrinth disorders) | 2/43
Hearing-Other (Ear and labyrinth disorders) | 3/43
Hypothyroidism (Endocrine disorders) | 1/43
Constipation (Gastrointestinal disorders) | 2/43
Diarrhea NOS (Gastrointestinal disorders) | 2/43
Dry mouth (Gastrointestinal disorders) | 26/43
Dysphagia (Gastrointestinal disorders) | 6/43
Esophageal spasm (Gastrointestinal disorders) | 1/43
Esophagitis NOS (Gastrointestinal disorders) | 6/43
GI-other (Gastrointestinal disorders) | 3/43
Gastric ulcer (Gastrointestinal disorders) | 1/43
Nausea (Gastrointestinal disorders) | 10/43
Radiation mucositis (Gastrointestinal disorders) | 14/43
Salivary gland disorder NOS (Gastrointestinal disorders) | 18/43
Stomatitis (Gastrointestinal disorders) | 3/43
Vomiting NOS (Gastrointestinal disorders) | 7/43
Chest pain (General disorders) | 1/43
Fatigue (General disorders) | 17/43
Infection NOS (General disorders) | 1/43
Late RT Toxicity: Esophagus (General disorders) | 4/38
Late RT Toxicity: Joint (General disorders) | 3/38
Late RT Toxicity: Larynx (General disorders) | 6/38
Late RT Toxicity: Mucous Membrane (General disorders) | 9/38
Late RT Toxicity: Other (General disorders) | 10/38
Late RT Toxicity: Salivary Gland (xerostomia, taste impairme (General disorders) | 22/38
Late RT Toxicity: Skin (within XRT field) (General disorders) | 6/38
Late RT Toxicity: Subcutaneous Tissue (Within XRT field) (General disorders) | 6/38
Pain due to radiation (General disorders) | 11/43
Pain-other (General disorders) | 8/43
Pyrexia (General disorders) | 2/43
Rigors (General disorders) | 1/43
Allergy-Other (Immune system disorders) | 1/43
Infection, Other (Infections and infestations) | 5/43
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 12/43
Blood creatinine increased (Investigations) | 1/43
Leukopenia NOS (Investigations) | 3/43
Weight decreased (Investigations) | 12/43
Anorexia (Metabolism and nutrition disorders) | 7/43
Blood albumin decreased (Metabolism and nutrition disorders) | 1/43
Blood magnesium decreased (Metabolism and nutrition disorders) | 1/43
Dehydration (Metabolism and nutrition disorders) | 5/43
Hypokalemia (Metabolism and nutrition disorders) | 1/43
Joint, muscle, or bone-Other (Musculoskeletal and connective tissue disorders) | 5/43
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 1/43
Depressed level of consciousness (Nervous system disorders) | 1/43
Peripheral motor neuropathy (Nervous system disorders) | 1/43
Peripheral sensory neuropathy (Nervous system disorders) | 1/43
Taste disturbance (Nervous system disorders) | 23/43
Anxiety NEC (Psychiatric disorders) | 2/43
Insomnia NEC (Psychiatric disorders) | 2/43
Sexual/reproductive function-Other (Reproductive system and breast disorders) | 1/43
Cough (Respiratory, thoracic and mediastinal disorders) | 5/43
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2/43
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 5/43
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2/43
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1/43
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 2/43
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 6/43
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1/43
Skin discoloration (Skin and subcutaneous tissue disorders) | 1/43
Skin-Other (Skin and subcutaneous tissue disorders) | 2/43
Acute Surgical Complication: Facial edema (Surgical and medical procedures) | 6
Acute Surgical Complication: Facial edema on the transfer si (Surgical and medical procedures) | 6
Acute Surgical Complication: Gland movement out of position (Surgical and medical procedures) | 1
Acute Surgical Complication: Neck numbness (Surgical and medical procedures) | 3
Acute Surgical Complication: Neck numbness on the transfer s (Surgical and medical procedures) | 2
Acute Surgical Complication: Nerve injury: hypoglossal (Surgical and medical procedures) | 1
Acute Surgical Complication: Nerve injury: hypoglossal on th (Surgical and medical procedures) | 1
Acute Surgical Complication: Nerve injury: lingual (Surgical and medical procedures) | 1
Acute Surgical Complication: Other (Surgical and medical procedures) | 4
Acute Surgical Complication: Shoulder weakness (Surgical and medical procedures) | 2
Acute Surgical Complication: Shoulder weakness on the transf (Surgical and medical procedures) | 1
Late Surgical Complication: Other (Surgical and medical procedures) | 10
Late Surgical Complication: Recurrent adenitis (Surgical and medical procedures) | 1
Late Surgical Complication: Submental fullness (Surgical and medical procedures) | 8
Edema NOS (Vascular disorders) | 3/43
Hemorrhage-Other (Vascular disorders) | 1/43
Lymphangiopathy NOS (Vascular disorders) | 2/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No